CLINICAL TRIAL: NCT02961699
Title: Healing Chronic Venous Stasis Wounds With Autologous Cell Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: InGeneron, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVSWH-001
Record Dates: First submitted 2016-11-09; First posted 2016-11-11 (Estimated); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Wound, Nonpenetrating
MeSH Terms: conditions — Wounds, Nonpenetrating | interventions — Debridement; Bandages

STUDY DESIGN:
Intervention Model Description: this study utilizes a medical device
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Transpose ® RT System (Experimental): Adipose-derived stem cells (also known as stromal vascular fraction or SVF) will be injected subcutaneously around the rim of the wound bed following standard would debridement. The standard collagen dressing material will also be saturated with SVF after placement within the would itself. Normal (standard) dressing of wound will be placed over wound.
  Interventions: Device: Transpose ® RT System
- debridement/dressing of wound (Active Comparator): Wound will be debrided and collagen dressing placed within wound bed as per standard of care. Standard dressing will cover wound. No adipose-derived stem cells (SVF) will be applied to control subject wounds.
  Interventions: Other: debridement/dressing of wound

INTERVENTIONS:
Device: Transpose ® RT System — adipose-derived stem cell therapy
  Arms: Transpose ® RT System
Other: debridement/dressing of wound — standard of care debridement and wound dressing
  Arms: debridement/dressing of wound

SUMMARY:
This is a prospective, randomized, single-site, safety and efficacy study of subjects with chronic venous stasis ulcers. Patients will fall into two categories: treatment arm (24 subjects) and non-treatment or control arm (12 subjects). The treatment group will undergo a small liposuction procedure and receive placement of autologous cell therapy (stromal vascular fraction or SVF) injected around the rim of venous stasis wound (subcutaneously)following standard wound debridement, with saturation of collagen dressing material with standard over-dressing. Control (non-treatment) subjects will receive debridement and dressing changes as per standard of care without SVF.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 years of age or older
* venous leg ulcers present for at least six months and not responding to
* standard wound therapy for at least one month prior to study treatment
* one wound size 10-25centimeters squared
* inpatient or outpatient treatment of chronic venous ulcers
* the ability of subjects to give appropriate consent or have an appropriate representative available

Exclusion Criteria:

* Age < 18 years of age
* Patients who are pregnant or currently breast feeding
* for a female subject of childbearing potential, a pregnancy test must be performed with negative results known within 7 days prior to the procedure
* Patient with a BMI less than or equal to 18.5 or an insufficient amount of subcutaneous tissue to allow recovery of up to 100ml of lipoaspirate
* Patients with poor glucose metabolic control (HgbA1c > 9)
* history of local neoplasm and any history of local neoplasm and any history of local neoplasm at site of administration
* History of systemic malignant neoplasms within last 5 years
* Patients who require Negative Pressure Wound Therapy (NPWT) or limb amputation at the target wound at the time of screening
* Wounds which are unable to be staged or classified. For example, full thickness tissue loss in which actual depth of the ulcer is completely obscured by slough and/or eschar in the wound bed
* Wounds that have evidence of necrosis after debridement
* Severe vascular disease in the pathogenesis of the ulcer (ABI<0.6)
* Clinical signs of critical colonization or local infection
* Prolonged(>6 months) of use of steroids
* Patients on an active regimen of chemotherapy
* Patients who have received radiation in proximity of the wound
* Patients with a documented history of liver disease or an ALT value>400
* Allergy to sodium citrate of any "caine" type of local anesthetic
* Subject is in the opinion of the Investigator or designee, unable to comply with the requirements of the study protocol or is unsuitable for the study for any reason. This includes completion of the Patient Reported Outcome instruments.
* Subject is currently participating in another clinical trial that has not yet completed its primary endpoint.
* Subject is part of a vulnerable population who, in the judgement of the investigator, is unable to give Informed Consent for reasons of incapacity, immaturity, adverse personal circumstances or lack of autonomy. This may include: Individuals with mental disability, person in nursing homes, children, impoverished persons, persons in emergency situations, homeless person, nomads, refugees, and those incapable of giving informed consent. Vulnerable populations also may include members of a group with a hierarchical structure such as university students, subordinate hospital and laboratory personnel, employees of the Sponsor, members of the armed forces, and persons kept in detention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Safety: as indicated through adverse event rate between control versus experimental group | enrollment through 12 months of follow-up
  adverse event rate
Time to complete wound closure as evidenced by complete epithelialization over a one-year time period (efficacy) | enrollment through 12 months of follow-up
  time it takes for complete wound closure following procedure

SECONDARY OUTCOMES:
Change in wound area over time (wound healing velocity) | enrollment through 12 months of follow-up
  size of wound will become smaller as measured during follow-up visits
Percent decrease in wound size (length X width X depth) | enrollment through 12 months of follow-up
  wound size will decrease when measured at follow-up visits
Patient-reported outcomes are informational endpoints to assess Health-Related Quality of Life | enrollment through 12 months of follow-up
  patient will report better health outcomes using quality of life questionnaires
Assessment of overall health status (questionnaire 36-Item Short Form/SF-36) | enrollment through 12 months of follow-up
  patient will report better health outcomes using quality of life questionnaires
assessment of disease specific quality of life (questionnaire: CIVIQ-20) | enrollment through 12 months of follow-up
  quality of life as it relates to lower extremity wound will improve following treatment as noted in patient's CIVIQ-20 scores

CONTACTS AND LOCATIONS:
Overall Officials: Bradley K Coots, M.D., Principal Investigator — Sanford Plastic and Reconstructive Surgery- Sioux Falls, SD
Locations (1):
- Sanford USD Medical Center, Sioux Falls, South Dakota, United States

IPD SHARING:
Plan to Share IPD: No